CLINICAL TRIAL: NCT05999370
Title: Is Correction of Malnutrition Sufficient to Improve Low Physical Function Before Elective Colorectal Cancer Surgery? A Randomized Controlled Trial of Nutrition vs Nutrition and Exercise Prehabilitation
Brief Title: Prehabilitation for Colorectal Cancer Patients With Low Functional Capacity and Malnutrition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Chelsia Ann Gillis, Assistant Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37-2021-6990
Record Dates: First submitted 2023-07-12; First posted 2023-08-21 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Prehabilitation; Malnutrition; Physical Functional Performance
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrition and exercise (Other): The nutrition intervention will be based on a comprehensive nutrition assessment by a dietitian at baseline, enabling individualized caloric and protein targets.
  The exercise intervention will be personalized based on a comprehensive assessment to include both a resistance and an aerobic component in the form of a "snack".
  Interventions: Behavioral: Nutrition; Behavioral: Exercise
- Nutrition only (Other): The nutrition intervention will be based on a comprehensive nutrition assessment by a dietitian at baseline, enabling individualized caloric and protein targets.
  Interventions: Behavioral: Nutrition

INTERVENTIONS:
Behavioral: Nutrition — The nutrition intervention will be based on needs assessed by indirect calorimetry, patient-generated subjective global assessment, and 24hr recall conducted at baseline, enabling individualized caloric and protein targets.
  Deficits in nutrient intake will be addressed with one-on-one dietary counselling and supplementation at baseline in a quantity that matches the estimated deficit in intake. Adherence will be monitored using 24-hr recalls and weight status by the dietitian weekly.
Behavioral: Exercise — The exercise intervention will include both a resistance and an aerobic component to be performed a total of 5 times a day, 5 times per week, 5 minutes each session, totaling 125 minutes per week. The ability to perform exercises as prescribed will be monitored with a weekly in-person or virtual supervised session.
  Arms: Nutrition and exercise

SUMMARY:
Despite multi-modal prehabilitation (nutrition, exercise, and psychosocial interventions), 60% of older elective colorectal cancer surgery patients with poor physical function were unable to reach a minimum preoperative 400m six-minute walking distance (6MWD), a prognostic cut-point. Compared to the patients that attained >400m 6MWD preoperatively, twice as many of <400m patients were malnourished. Malnutrition has long been associated with worse functioning (e.g., physical, immune). The investigators hypothesize that for nutritionally deficient patients, the etiology for their poor physical function is malnutrition. Correction of malnutrition alone might thus be sufficient to achieve a 400m 6MWD before surgery and improve patient outcomes.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled trial of nutrition prehabilitation alone vs nutrition prehabilitation with supportive exercise in patients with malnutrition and 6MWD <400m before elective colorectal surgery. The primary objective, and therapeutic target, will be achievement of minimal clinical important difference for the 6MWD (14m for within group comparisons and 19m between groups). Ability to adhere to the interventions will be monitored. The findings of this study will guide optimal treatment for this vulnerable population by exploring the role of nutrition alone vs. nutrition with exercise to optimize surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older;
* Patients with cancer scheduled for primary colorectal resection;
* Patients with 6MWD at baseline less than 400 m;
* Patients with Patient-Generated Subjective-Global Assessment (malnutrition assessment) score equal or greater than 9.

Exclusion Criteria:

* Patients with history of premorbid conditions that contraindicate exercise including dementia, -Parkinson's disease or previous stroke with paresis;
* Metastatic cancer;
* Patients who do not speak English or French and cannot be accompanied by someone who speaks English or French;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Preoperative six-minute walking distance | from date of baseline assessment until date of surgery, an average of 4 weeks, recorded in meters
  Physical function will be measured with the six-minute walking test (6MWT). Patients will be instructed to walk back and forth along a 20m hallway, and the distance covered in 6 minutes (6MWD) will be recorded (meters).

SECONDARY OUTCOMES:
Adherence to the exercise intervention | from date of baseline assessment until date of surgery,an average of 4 weeks, recorded in steps
  Adherence will be monitored by use of logbooks and a smart watch (FitBit), which records daily steps.
Adherence to the nutrition intervention | from date of baseline assessment until date of surgery, an average of 4 weeks, recorded in % of prescription adherence
  Adherence to dietary targets (energy intake) will be carefully monitored by weekly in-person or virtual visit using 24hr recalls and supplement counts (energy consumption as compared to prescribed energy targets)
Adherence to the nutrition intervention | from date of baseline assessment until date of surgery, an average of 4 weeks, recorded in % of prescription adherence
  Adherence to dietary targets (protein intake) will be carefully monitored by weekly in-person or virtual visit using 24hr recalls and supplement counts (protein consumption as compared to prescribed protein targets)

CONTACTS AND LOCATIONS:
Overall Officials: Chelsia Gillis, RD PhD, Principal Investigator — McGill University
Locations (1):
- MUHC Research Ethics Board, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillis C, Fenton TR, Gramlich L, Keller H, Sajobi TT, Culos-Reed SN, Richer L, Awasthi R, Carli F. Malnutrition modifies the response to multimodal prehabilitation: a pooled analysis of prehabilitation trials. Appl Physiol Nutr Metab. 2022 Feb;47(2):141-150. doi: 10.1139/apnm-2021-0299. Epub 2021 Sep 29. PMID 34587460
- [Background] Carli F, Bousquet-Dion G, Awasthi R, Elsherbini N, Liberman S, Boutros M, Stein B, Charlebois P, Ghitulescu G, Morin N, Jagoe T, Scheede-Bergdahl C, Minnella EM, Fiore JF Jr. Effect of Multimodal Prehabilitation vs Postoperative Rehabilitation on 30-Day Postoperative Complications for Frail Patients Undergoing Resection of Colorectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Mar 1;155(3):233-242. doi: 10.1001/jamasurg.2019.5474. PMID 31968063
- [Background] Gillis C, Buhler K, Bresee L, Carli F, Gramlich L, Culos-Reed N, Sajobi TT, Fenton TR. Effects of Nutritional Prehabilitation, With and Without Exercise, on Outcomes of Patients Who Undergo Colorectal Surgery: A Systematic Review and Meta-analysis. Gastroenterology. 2018 Aug;155(2):391-410.e4. doi: 10.1053/j.gastro.2018.05.012. Epub 2018 May 8. PMID 29750973
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Background] Gillis C, Fenton TR, Gramlich L, Sajobi TT, Culos-Reed SN, Bousquet-Dion G, Elsherbini N, Fiore JF Jr, Minnella EM, Awasthi R, Liberman AS, Boutros M, Carli F. Older frail prehabilitated patients who cannot attain a 400 m 6-min walking distance before colorectal surgery suffer more postoperative complications. Eur J Surg Oncol. 2021 Apr;47(4):874-881. doi: 10.1016/j.ejso.2020.09.041. Epub 2020 Oct 5. PMID 33041092